CLINICAL TRIAL: NCT03031808
Title: Comparison of Two Induction Regimens Using Topical Lidocaine or Muscle Relaxant; Impact on Postoperative Sore Throat and Haemodynamics
Brief Title: Comparison of Two Induction Regimens Using Topical Lidocaine or Muscle Relaxant on Sore Throat and Hemodynamics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Jan Sverre Vamnes, Senior consultant, Ph.D., Ostfold Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB3383
Record Dates: First submitted 2016-12-21; First posted 2017-01-26 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Intubation Complication
MeSH Terms: interventions — Rocuronium; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine spray (Other): Endotracheal lidocaine spray prior to intubation
  Interventions: Drug: Lidocaine spray (2%)
- Muscle relaxant (Other): Muscle relaxant prior to intubation
  Interventions: Drug: Muscle Relaxant (Rocuronium)
- No Muscle relaxant, no Lidocaine (Other): 'No Muscle relaxant, no Lidocaine Control group
  Interventions: Other: No Muscle relaxant, no Lidocaine

INTERVENTIONS:
Drug: Lidocaine spray (2%) — Spraying trachea from 2 cm above the vocal cords and 5 cm down with a straw with multiple side holes
  Other Names: Xylocain 2% Astra Zeneca
  Arms: Lidocaine spray
Drug: Muscle Relaxant (Rocuronium) — After induction of anesthesia, the participants are given 0,6 mg/kg bodyweight intravenously.
  Other Names: Esmeron MSD
  Arms: Muscle relaxant
Other: No Muscle relaxant, no Lidocaine — This group get general anesthesia without Rocuronium or Lidocaine
  Other Names: Control group
  Arms: No Muscle relaxant, no Lidocaine

SUMMARY:
When a surgical procedure is performed under general anesthesia, the Airways are often secured With an endotracheal tube. Some patients experience sore throat thereafter. Studies have shown a reduction of these side effects when by use of muscle relaxants or a lidocain spray prior to the intubation. At Ostfold Hospital Trust, the investigators use one of the two methods or nothing. These methods will be studied systematically.

Heart rate and blood pressure rise during the intubation procedure. The investigators will also study the differences between the groups.

DETAILED DESCRIPTION:
Post-operative sore throat and cough are common complications of endotracheal intubation and occurs in 30% to 70% of patients. Spraying with Lidocaine reduces this incident of postoperative sore Throat (POST). The use of neuromuscular blocking agents (NMBA) alone will also diminish the incidence of adverse postoperative upper airway symptoms. The use of topical Lidocaine is shown to reduce the cardiovascular responses during and after endotracheal intubation.

Hypertension and tachycardia as a response to endotracheal intubation are probably of little consequence in healthy individuals. These reactions might though be harmful in patients with cardiovascular diseases.

Postoperative sore throat is an undesired outcome for the patient. Topical or systemic pharmacological interventions is shown to reduce the POST.

Our anesthetists practice very different. The investigators sometime use topical lidocaine 2% as a spray, sometime muscle relaxants and often nothing but propofol and remifentanil prior to laryngoscopy an endotracheal intubation.

The objective of this study is to determine, whether the use of topical administered lidocaine, 2 %, has a better impact on POST compared with NMBA alone in general anesthesia with propofol and remifentanil. Patients receiving nothing but propofol and remifentanil will be the reference group. Assessment of the intubation conditions will be done according to a standard scheme

The primary endpoint:

* Differences in the intubation conditions between the three groups.
* Cardiovascular responses caused by the laryngoscopy and intubation.

The secondary endpoint:

• Post operative upper airways symptoms. Power and Sample Size Calculator To detect a decrease in the incidence of pharyngolaryngeal symptoms from 60% to 45%, we calculated that we needed 150 patients per study arm (power of the study, 0,8; type I error, 0,05).

450 adult patients have to be scheduled for the study.

The study is double blind, randomized:

* Group Topical lidocaine 4%:
* Group NMBA
* Control group Premedication: Paracetamol 2g General anaesthesia: TCI (Target Control of Infusion is a principle, an anesthesia infusion after protocol): Propofol and Remifentanil Surgical procedure: Not specified short lasting (<1 h) procedures The experienced anesthesiologist performing the intubating procedure will not be in the room until immediately before the intubation.

Postoperatively:

* Oral paracetamol and codeine-fixed combination up to 1000 mg and 60 mg, respectively, every 6 h
* When nausea and vomiting occurs postoperatively, ondansetron 4 mg IV administers as the drug of first choice followed by droperidol 0,625 mg IV if the nausea/vomiting persists.

Collected data:

* Patient characteristics inclusive smoke habits
* Intubation conditions according to the Copenhagen score
* Blood pressure prior to laryngoscopy and after 1, 3, 5, 7, 9, 11, 13 and 15 minutes, then every 15 min.
* Cuff pressure
* Pharyngolaryngeal discomfort 2 and 24 hours (telephone interview if released from hospital) after extubation

ELIGIBILITY:
Inclusion Criteria:

* Scheduled elective surgery with general anesthesia and planned endotracheal intubation.

Exclusion Criteria:

* ASA≥3,
* 20>BMI<35
* Allergy to local anesthetics or neuromuscular blocking agents.
* The ASA physical status classification system is a system for assessing the fitness of patients before surgery. BMI is Body Mass Index measured in kilograms/square meter.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Sore Throat postoperative. Assessment of complaints and changes in complaints | 2 h and 24 h after extubation
  Postoperative sore throat, described 2 h and 24 h after extubation. If the patient has sore throat or is hoarse, the complaint is assessed on a VAS (Visual Analogue Scale) 1 - 10.
Intubation conditions directly after induction of anesthesia | 90 sec. after established general anesthesia
  Describes the intubation conditions: Jaw relaxation, resistance to laryngoscopy blade, the position and movement of vocal cords, the movement of limbs and coughing. Each variable rates as excellent, good or poor. Intubation conditions are many variables described once and should not be divided into several outcomes.
Hemodynamic parameters, change in HR (Heart Rate) is being assessed | Prior to induction, then every second minute the next 15 minutes, thereafter every 15 minute until end of surgery (max. 2 h.)
  Describes changes in HR (Heart Rate)
Hemodynamic parameters, change in BP (blood pressure) is being assessed | Prior to induction, then every second minute the next 15 minutes, thereafter every 15 minute until end of surgery (max. 2 h.)
  Describes changes in BP(Blood Pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sverre Vamnes, MD, Ph.D., Study Chair — Senior consultant
Locations (1):
- Ostfold Hospital Trust, Moss, Grålum, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: No
No sharing plan so far.

REFERENCES:
- [Background] Banihashem N, Alijanpour E, Hasannasab B, Zarei A. Prophylactic Effects of Lidocaine or Beclomethasone Spray on Post-Operative Sore Throat and Cough after Orotracheal Intubation. Iran J Otorhinolaryngol. 2015 May;27(80):179-84. PMID 26082898
- [Background] Blobner M, Mirakhur RK, Wierda JM, Wright PM, Olkkola KT, Debaene B, Pendeville P, Engbaek J, Rietbergen H, Sparr HJ. Rapacuronium 2.0 or 2.5 mg kg-1 for rapid-sequence induction: comparison with succinylcholine 1.0 mg kg-1. Br J Anaesth. 2000 Nov;85(5):724-31. doi: 10.1093/bja/85.5.724. PMID 11094588
- [Background] Combes X, Andriamifidy L, Dufresne E, Suen P, Sauvat S, Scherrer E, Feiss P, Marty J, Duvaldestin P. Comparison of two induction regimens using or not using muscle relaxant: impact on postoperative upper airway discomfort. Br J Anaesth. 2007 Aug;99(2):276-81. doi: 10.1093/bja/aem147. Epub 2007 Jun 15. PMID 17573390
- [Background] Domaoal AM, Weniger FC, Wolfson B. "Precurarization" using pancuronium. Anesth Analg. 1975 Jan-Feb;54(1):71-5. doi: 10.1213/00000539-197501000-00014. PMID 1167764
- [Background] Doyle DJ. Airway anesthesia: theory and practice. Anesthesiol Clin. 2015 Jun;33(2):291-304. doi: 10.1016/j.anclin.2015.02.013. PMID 25999003
- [Background] Kalil DM, Silvestro LS, Austin PN. Novel preoperative pharmacologic methods of preventing postoperative sore throat due to tracheal intubation. AANA J. 2014 Jun;82(3):188-97. PMID 25109156
- [Background] Martin C, Bonneru JJ, Brun JP, Albanese J, Gouin F. Vecuronium or suxamethonium for rapid sequence intubation: which is better? Br J Anaesth. 1987 Oct;59(10):1240-4. doi: 10.1093/bja/59.10.1240. PMID 2890365
- [Background] Mostafa SM, Murthy BV, Barrett PJ, McHugh P. Comparison of the effects of topical lignocaine spray applied before or after induction of anaesthesia on the pressor response to direct laryngoscopy and intubation. Eur J Anaesthesiol. 1999 Jan;16(1):7-10. doi: 10.1046/j.1365-2346.1999.00410.x. PMID 10084094
- [Background] Koller ME, Husby P. High-dose vecuronium may be an alternative to suxamethonium for rapid-sequence intubation. Acta Anaesthesiol Scand. 1993 Jul;37(5):465-8. doi: 10.1111/j.1399-6576.1993.tb03747.x. PMID 7741805
- [Background] Qi DY, Wang K, Zhang H, Du BX, Xu FY, Wang L, Zou Z, Shi XY. Efficacy of intravenous lidocaine versus placebo on attenuating cardiovascular response to laryngoscopy and tracheal intubation: a systematic review of randomized controlled trials. Minerva Anestesiol. 2013 Dec;79(12):1423-35. Epub 2013 Jul 9. PMID 23839320
- [Background] Tanaka Y, Nakayama T, Nishimori M, Sato Y, Furuya H. Lidocaine for preventing postoperative sore throat. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD004081. doi: 10.1002/14651858.CD004081.pub2. PMID 19588349
- [Background] Viby-Mogensen J, Engbaek J, Eriksson LI, Gramstad L, Jensen E, Jensen FS, Koscielniak-Nielsen Z, Skovgaard LT, Ostergaard D. Good clinical research practice (GCRP) in pharmacodynamic studies of neuromuscular blocking agents. Acta Anaesthesiol Scand. 1996 Jan;40(1):59-74. doi: 10.1111/j.1399-6576.1996.tb04389.x. PMID 8904261